CLINICAL TRIAL: NCT03719768
Title: Phase IB Study of Avelumab With Radiotherapy in Patients With Leptomeningeal Disease
Brief Title: Avelumab With Radiotherapy in Patients With Leptomeningeal Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19648; W1239387 (Other: Pfizer)
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Leptomeningeal Metastases; Leptomeningeal Disease
Keywords: Whole Brain Radiotherapy; meningeal; LMDz; brain metastases; Immunotherapy
MeSH Terms: conditions — Meningeal Carcinomatosis; Meningeal Neoplasms; Brain Neoplasms | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avelumab and Whole Brain Radiotherapy (Experimental): Avelumab 800 mg intravenously (IV) and 3000 centriGray units (cGy) Whole Brain Radiotherapy once every 2 weeks
  Interventions: Drug: Avelumab; Radiation: Whole Brain Radiotherapy

INTERVENTIONS:
Drug: Avelumab — Patients will be given 800 mg Avelumab as a one hour intravenous infusion once every 2 weeks.
  Other Names: Bavencio
Radiation: Whole Brain Radiotherapy — Patients will be given 3000 cGy Whole Brain Radiotherapy once every 2 weeks
  Other Names: WBRT

SUMMARY:
This study is to find a safe dose of the combination of Avelumab and Whole Brain Radiotherapy (WBRT) in patients with Leptomeningeal Disease.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically or cytologically confirmed diagnosis of any cancer except leukemia
* 2. Patients must have the presence of malignant cells in the CSF (CSF+) OR at least 2 of the 3 following features: 1) clinical signs and symptoms of LMDz 2) characteristic radiographic abnormalities , and 3) "suspicious" CSF (Chamberlain 2017)
* 3. Patients must have an Eastern Cooperative Oncology Group performance scale of < 3 OR Karnofsky Performance Status of >50.
* 4. An interval of at least 2 weeks after the end of prior radiation therapy to the brain (e.g., stereotactic radiosurgery or other-WBRT is excluded)
* 5. An interval of at least 4 weeks following any surgical resection of brain lesions prior to treatment
* 6. Be > 18 years of age on the day of signing consent
* 7. Demonstrate adequate organ function as defined in Table 2. All screening labs should be performed with 14 days of treatment initiation
* 8. Resting baseline O2 saturation by pulse oximetry of > 92% at rest
* 9. Patients must have recovered from the toxic effects of prior therapies (< Grade 1)
* 10. Provision of signed and dated informed consent form
* 11. Life expectancy of > 8 weeks
* 12. Pregnancy test: negative serum or urine pregnancy test at screening for women of childbearing potential.
* 13. Contraception: Highly effective contraception for both male and female subjects throughout the study and for at least 30 days after last Avelumab treatment administration, if the risk of conception exists.
* 14. If the disease has progressed on current treatment in the CNS prior to consent, patients may continue Her 2 directed antibody treatment (trastuzumab and pertuzumab), aromatase inhibitor or tamoxifen while on the study; patients with triple negative breast cancer may continue capecitabine, eribulin or paclitaxel while on the study per PI discretion.
* 15. Adequate Organ Function as defined per protocol

Exclusion Criteria:

* 1. Receiving other treatments specifically administered to treat LMDz or antibody based therapies within the last 4 weeks. However, patients receiving concomitant non-cytotoxic therapy (hormonal or cytostatic therapy) to control systemic disease or bulk CNS disease will be eligible, provided the therapy is not a phase I agent, an agent which significantly penetrates the CSF (e.g., high-dose methotrexate, thiotepa, or high-dose ara-C), or an agent known to have serious unpredictable CNS side effects Except as listed in Inclusion Criteria #15 (above). Careful documentation of concurrently administered systemic drugs is required
* 2. Patients with a ventriculoperitoneal or ventriculoatrial shunt must have an on/off device in their shunt systems to be eligible for the study. Patients must be able to tolerate shunt closure for ~4 hours without development of clinical signs of increased intracranial pressure. Patients unable to tolerate shunt closure for ~4 hours will not be eligible for the study
* 3. Unable or unwilling to have a contrast-enhanced brain MRI
* 4. Currently participating in or having participated in a study of an investigational agent or device < 4 weeks prior to the first dose of study treatment
* 5. Patients on steroid therapy unless < 2 mg/day dexamethasone equivalents
* 6. Prior chemotherapy or targeted small molecule therapy except as listed in Inclusion Criteria #15 and Exclusion #1(above) within 4 weeks prior to study Day 1 or nonrecovery (i.e., < Grade 1 or at baseline) from adverse events (AEs) due to agents administered > 4 weeks earlier
* 7. Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* 8. Has an active autoimmune disease requiring systemic treatment within the past 3 months (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive agents) or has a diagnosis of immunodeficiency. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study. Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* 9. Has evidence of active, non-infectious pneumonitis
* 10. Has an active infection requiring systemic therapy
* 11. Had major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 1 of treatment on study. Ommaya placement is allowed
* 12. Requires escalating or chronic supraphysiologic doses of corticosteroids (> 10 mg/day prednisone equivalents)
* 13. Has a history of current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* 14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* 15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 90 days after the last dose of trial treatment
* 16. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti- Cytotoxic T-lymphocyte-associated antigen-4 (cTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways) within 6 months before the beginning of study treatment
* 17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1, 2 antibodies)
* 18. Any test for hepatitis B (HBV) or hepatitis C virus (HCV) indicating acute or chronic infection
* 19. Has received a live vaccine within 30 days prior to the first dose of trial treatment
* 20. Prior administration of WBRT
* 21. Known symptomatic brain metastases requiring steroids. Patients with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to study treatment, have discontinued corticosteroid treatment for these metastases for at least 4 weeks and are neurologically stable. Short courses of corticosteroids are permitted if these were started for leptomeningeal disease and can be tapered down to < 2 mg/day of dexamethasone equivalents and patients remain stable for 3 days prior to study treatment
* 22. Known severe hypersensitivity reactions to monoclonal antibodies (Grade > 3) or any known history of anaphylaxis
* 23. ORGAN TRANSPLANTATION: Prior organ transplantation including allogenic stem-cell transplantation
* 24. CARDIOVASCULAR DISEASE: Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (> New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication
* 25. OTHER PERSISTING TOXICITIES: "Persisting toxicity related to prior therapy (NCI CTCAE v.5.0 Grade > 1); however, alopecia, sensory neuropathy Grade < 2, or other Grade < 2 not constituting a safety risk based on investigator's judgment are acceptable
* 26. Other severe acute or chronic medical conditions, including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Safety and Dose Limiting Toxicity (DLT) measured by number of subjects with adverse events (AEs) | End of treatment (3 months)
  Adverse events will only include those that are determined to be related to study drug.
  A DLT will be defined as any one of the following adverse events occurring within 28 days from first dose of Avelumab. Central Nervous System (CNS) toxicities: Any grade 3 or higher central nervous adverse events, including but not limited to cerebral hemorrhage and new-onset neurologic deficit. Non-CNS toxicities: Any grade 3 or higher nonhematologic AE with the exception of alopecia and fatigue - Grade > 3 nausea, vomiting, or diarrhea despite maximal medical therapy - Grade > 3 laboratory value if 1)medical intervention is required to treat the patient or 2) the abnormality leads to hospitalization • Any grade 3 or 4 event that does not improve within 6 weeks

SECONDARY OUTCOMES:
Number of T Cells | Up to 11 months
  The number of T cells in the cerebrospinal fluid (CSF) and the CSF cytokine activation profile in the CSF (relative to serum) measured before and after Avelumab administration.
Activation Status of T Cells | Up to 11 months
  The activation status of T cells in the cerebrospinal fluid (CSF) and the CSF cytokine activation profile in the CSF (relative to serum) measured before and after Avelumab administration.

OTHER OUTCOMES:
Overall Survival (OS) Rate at 3 months | 3 months
  OS, utilizing 95% confidence interval (95%CI).

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Forsyth, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Pina Y, Law V, Sahebjam S, Tran N, Siddarajappa N, Li J, Mo Q, Phadke MS, Arrington J, Macaulay R, Mokhtari S, Evernden B, Ahmed KA, Smalley I, Yu M, Smalley KSM, Forsyth PA. Phase IB Study of Avelumab and Whole Brain Radiotherapy (WBRT) in Patients with Leptomeningeal Disease (LMD) from Solid Tumors: Results and Molecular Analyses. Neuro Oncol. 2025 Aug 28:noaf183. doi: 10.1093/neuonc/noaf183. Online ahead of print. PMID 40888040